CLINICAL TRIAL: NCT06912542
Title: GLYCEMIC RESPONSE AFTER CONSUMPTION OF FRENCH BREAD WITH WHOLE OR GROUND FLAXSEEDS IN PEOPLE WITH TYPE 2 DIABETES MELLITUS
Brief Title: ACUTE EFFECT OF CONSUMPTION OF GROUND OR WHOLE FLAXSEEDS ON BLOOD GLUCOSE IN PEOPLE WITH TYPE 2 DIABETES
Acronym: DM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Francisca (Other)
Collaborators: Universidade Franciscana (UFN)- Brasil (Unknown)
Responsible Party: Principal Investigator, Laureana Q Barcelos, Mestre em Ciências da Saúde e da Vida, Universidade Francisca
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 5.747.049; 64777622.00000.5306 (Registry Identifier: CAAE - Certificate of Presentation of Ethical Appreciation); Research Ethics Committee (Registry Identifier: 5.747.049)
Record Dates: First submitted 2025-03-10; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Diabetes; Diabetes Type 2; Insulin Resistance
Keywords: Postprandial Period; Glycemic Control; Flax; Bread
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Randomized, crossover clinical study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Whole flaxseed bread (Active Comparator): The 16 participants consumed 1 serving of bread with 30 g of whole flaxseeds in one of the three study interventions.
  Interventions: Other: Whole flaxseed bread
- Bread with ground flaxseed (Active Comparator): The 16 participants consumed 1 serving of bread with 30 g of ground flaxseeds in one of the three study interventions.
  Interventions: Other: Ground flaxseed bread
- Control bread (Placebo Comparator): The 16 participants consumed 1 serving of control bread (without flaxseeds) in one of the three study interventions.
  Interventions: Other: French bread

INTERVENTIONS:
Other: Whole flaxseed bread — French bread with the addition of 30g of whole flaxseed.
  Arms: Whole flaxseed bread
Other: Ground flaxseed bread — French bread with the addition of 30g of ground flaxseed.
  Arms: Bread with ground flaxseed
Other: French bread — Plain French bread (control).
  Arms: Control bread

SUMMARY:
This study aimed to evaluate the effect of consuming a portion of French bread combined with whole or ground flaxseed on the glycemia of people with DM 2 in a randomized, crossover clinical trial conducted with 16 people with DM 2 who were not using insulin.

The main questions of the study were:

1. Is flaxseed able to control the glycemia of people with type 2 diabetes?
2. What is the best way to consume flaxseed to control the glycemia of people with type 2 diabetes?

The 3 types of bread (whole flaxseed, ground flaxseed and control) were evaluated in interventions, with a 7-day interval between them, for the consumption of the bread and evaluation of the behavior of the glycemia and insulin curve.

DETAILED DESCRIPTION:
This study aimed to evaluate the effect of consuming a portion of French bread combined with whole or ground flaxseed on the blood glucose levels of people with DM 2 in a randomized, crossover clinical trial conducted with 16 people with DM 2 who were not taking insulin.

The main questions of the study were:

1. Is flaxseed able to control the blood glucose levels of people with type 2 diabetes?
2. What is the best way to consume flaxseed to control the blood glucose levels of people with type 2 diabetes? People with type 2 diabetes mellitus participated in the study, divided into three groups for random consumption of the breads: French bread without flaxseed (control bread), French bread with 30g of whole flaxseed, and French bread with 30g of ground flaxseed. The design was crossover and had a 7-day washout. Capillary blood glucose levels were monitored during fasting and at 15, 30, 60, 90 and 120 minutes after ingestion of the breads, while serum glucose and insulin levels were measured during fasting and at peak blood glucose levels, at 60 minutes. In addition, sociodemographic and clinical data (medication use, duration of DM2, bowel habits, sleep, and physical activity), nutritional status, and pre-intervention food consumption with a 24-hour dietary recall were evaluated. The data were analyzed in the R statistical software, through the Shapiro-Wilk normality test, one-way ANOVA, with Tukey or Kruskal-Wallis post-hoc. The analyses had a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* The selection included individuals with DM 2
* Of both sexes
* Adults and elderly individuals without risk of dysphagia
* Aged 18 years or older
* Without allergies to the test foods
* With the habit of having breakfast (≥4 days a week, with an intake of ≥100 kcal within two hours of waking up)
* Availability of time for the days planned for the research.

Exclusion Criteria:

* The exclusion criteria were applied to individuals diagnosed with another type of Diabetes
* Using exogenous insulin
* Pregnant or lactating women
* Smokers
* With diseases that affect taste
* The gastrointestinal system, and who reported the last intestinal frequency according to the Bristol scale 1, 2, 5, 6 and 7.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose concentration | In the 3 interventions, completed in 3 weeks.
  Six capillary blood glucose tests were performed in each study intervention. Time 0 (zero) was the basal measurement, and the others were performed in the postprandial period at 15, 30, 90 and 120 minutes.

SECONDARY OUTCOMES:
Insulin Concentration | In the 3 interventions, completed in 3 weeks.
  Two plasma insulin tests were performed in each study intervention. Time 0 (zero) was the basal measurement, and the other was at the peak of the postprandial period, considered at 60 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Laureana de Quevedo Barcelos, Mestre, Principal Investigator — Universidade Franciscana
Locations (1):
- Universidade Franciscana, Santa Maria, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Protocolo de estudo
Supporting Information: Study Protocol, ICF
Time Frame: Starting 1 year after publication with no end date.